CLINICAL TRIAL: NCT03062345
Title: Multi-user Virtual Training for Upper Extremity in the Home
Brief Title: In Home VR Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, James Patton, Co-Director, Robotics Laboratory, Sensory Motor Performance Program, Rehabilitation Institute of Chicago, Shirley Ryan AbilityLab
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: STU00204187
Record Dates: First submitted 2017-02-19; First posted 2017-02-23 (Actual); Last update posted 2021-06-10 (Actual); Status verified 2021-06

CONDITIONS: Stroke
Keywords: Stroke; Virtual Reality Therapy; Rehabilitation; Upper Extremity; Arm; Telerehabilitation
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-User Mode first, Multi-User Mode second (Experimental)
  Interventions: Other: Single-User Virtual Reality Upper Extremity Therapy; Other: Multi-User Virtual Reality Upper Extremity Therapy
- Multi-User Mode first, Single-User Mode second (Experimental)
  Interventions: Other: Single-User Virtual Reality Upper Extremity Therapy; Other: Multi-User Virtual Reality Upper Extremity Therapy

INTERVENTIONS:
Other: Single-User Virtual Reality Upper Extremity Therapy — Virtual Reality games with the user as the only person required for participation
  Other Names: Single-User Mode; Single-User Mode first, Multi-User Mode second; Multi-User Mode first, Single-User Mode second
Other: Multi-User Virtual Reality Upper Extremity Therapy — Virtual reality games in which more than one user is required for participation. Users interact in the virtual environment.
  Other Names: Multi-User Mode; Single-User Mode first, Multi-User Mode second; Multi-User Mode first, Single-User Mode second

SUMMARY:
Virtual reality is a video game in which a person and their real-time movements are represented on a screen in a virtual environment. This study will compare the use of multi-user virtual reality (VR) to single-user VR to determine if either provides superior engagement in upper extremity therapy and greater motivation to perform repetitive training.

Stroke survivors will participate in a longitudinal study in which they will have the opportunity to perform rehabilitative training with multi-user VR and single-user VR modes in their homes. They will use each mode for 2 weeks, completing 4 session per week, each session is 1 hour long. Upper extremity motor control, level of engagement, and active range of motion will be assessed at time points during the intervention period.

Subject evaluations will take place before the intervention, at the midpoint of intervention (between switching from multi-user to single-user modes, or vice versa), and at the end of the intervention.

The investigators hope to address two aims:

Aim 1: To determine if the use in-home multi-user virtual reality treatment results in greater engagement in therapy compared with in-home single user virtual reality treatment.

Aim 2: To determine if in-home virtual reality treatment results in greater practice

The investigators hypothesize that stroke survivors will be more engaged in therapy when training with the multi-user VR system and this will translate into greater practice.

ELIGIBILITY:
Inclusion Criteria:

* Are between the ages of 21 and 80
* Experienced a single stroke at least 6 months prior to enrollment
* Have moderate arm impairment as indicated by a score between 4 and 6 on the Chedoke-McMaster Stroke Assessment, arm subscale
* Live within 20 miles of the Rehabilitation Institute of Chicago (as study personnel will need to travel to their home)

Exclusion Criteria:

* Other neurological, neuromuscular, or orthopedic disease
* Pain in the upper extremity with movements required in the treatment
* Contracture that limits use of the VR system
* Vision problems which would preclude the ability to use the VR system
* Cognitive or language deficits that would prevent them from understanding the tasks
* Concurrent enrollment in another intervention study involving the affected arm or hand
* Botox injection in the arm within the previous 6 months

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2017-01-26 (Actual); Primary Completion 2018-05-31 (Actual); Study Completion 2020-05-30 (Actual)

PRIMARY OUTCOMES:
Hand displacement during each session | Distance hand moves on average per session during each 2-week treatment phase (each subject will complete 2, 2-week phases of treatment. One 2-week phase being the Single-user mode and the other 2-week phase being the Multi-user mode)
  total distance hand moves during all therapy sessions divided by the number of sessions in which a subject participates.

SECONDARY OUTCOMES:
Therapy mode amount of use | 2 week treatment phase
  Total amount of time subject spends in their assigned therapy mode during the 2-week treatment phase.
Change in Active Range of Motion | First measure taken at baseline, then also at the end of the first 2-week treatment phase and finally at the end of the second 2-week treatment phase.
  Change from baseline in angle of upper extremity movement (shoulder and elbow)
Comparison of Intrinsic Motivation Inventory Score between therapy modes | First measure taken at the end of the first 2-week treatment phase; Second measure taken at the end of the second 2-week treatment phase.
  Difference in Intrinsic Motivation Inventory score between single-user and multi-user modes

CONTACTS AND LOCATIONS:
Overall Officials: James Patton, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Thielbar KO, Triandafilou KM, Barry AJ, Yuan N, Nishimoto A, Johnson J, Stoykov ME, Tsoupikova D, Kamper DG. Home-based Upper Extremity Stroke Therapy Using a Multiuser Virtual Reality Environment: A Randomized Trial. Arch Phys Med Rehabil. 2020 Feb;101(2):196-203. doi: 10.1016/j.apmr.2019.10.182. Epub 2019 Nov 9. PMID 31715140